CLINICAL TRIAL: NCT03595540
Title: Phase II Clinical Study of a Fasting-mimicking Diet in Patients Undergoing Oncologic Treatment
Brief Title: Fasting-mimicking Diet in Patients Undergoing Active Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Alessio Nencioni, Associate Professor, University of Genova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 308CER2017
Record Dates: First submitted 2018-07-12; First posted 2018-07-23 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Cancer; Breast Cancer; Colorectal Cancer
Keywords: fasting-mimicking diet; cancer; nutritional status; body composition; fasting
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Fasting | interventions — Gestyl

STUDY DESIGN:
Intervention Model Description: This is a pilot, single arm prospective trial assessing feasibility and safety of a 5-day fasting-mimicking diet in patients with different cancer types and concomitant anticancer treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prolon - FMD (Experimental): Patients undergoing active cancer treatment are assigned monthly cycles of the fasting-mimicking diet Prolon
  Interventions: Other: Prolon

INTERVENTIONS:
Other: Prolon — Prolon by L-Nutra is a medically-designed dietary kit providing the food to eat for five days. Day 1 of Prolon provides ~4600 kJ (11% protein, 46% fat, and 43% carbohydrate), whereas days 2-to-5 provide ~3000 kJ (9% protein, 44% fat, and 47% carbohydrate) per day.
  Other Names: fasting-mimicking diet

SUMMARY:
This is a pilot, single arm prospective trial assessing feasibility, safety and effects on patient nutritional status of a 5-day fasting-mimicking diet (FMD) in patients with different cancer types and concomitant anticancer treatment.

DETAILED DESCRIPTION:
It is proposed to conduct a single-arm phase II clinical study of a FMD (Prolon, by L-Nutra) in 60 patients with solid or hematologic tumors who undergo treatment with chemotherapeutic regimens, hormone therapies, other molecularly targeted therapies (including kinase inhibitors), biological drugs (including trastuzumab, pertuzumab, cetuximab and bevacizumab) or inhibitors of immune checkpoints (e.g. Opdivo, Keytruda).

Prolon is a FMD lasting five days. It consist of vegetable soups, broths, bars, olives, crackers, herbal teas, supplements of vitamins and minerals. Day 1 of the FMD supplies ~4600 kJ (11% protein, 46% fat, and 43% carbohydrate), whereas days 2-to-5 provide ~3000 kJ (9% protein, 44% fat, and 47% carbohydrate) per day.

Primary endpoints of the study are the feasibility and safety of monthly cycles of the FMD in patients with solid or hematologic tumors who undergo active treatment. Feasibility is monitored through the compilation of a food diary and is defined as the strict adherence to the diet prescribed in all its days with the possibility of admitting the consumption of only 50% of the planned diet and / or a maximum consumption of 4-5 Kcal / kg body weight of food not provided in only one of the five days of each cycle. Furthermore, the dosage of IGF-1 and of urinary ketone bodies allow to identify further cases of non-adherence to the diet.

FMD-emergent side effects are monitored according to the NCI-CTCAE version 5.0.

Secondary endpoints include:

* patient nutritional status as monitored by weight, handgrip strength, bio-impedance and serum markers (ferritin, transferrin, colinesterase).
* Quality of life (QLQ-C30)
* Clinical responses measured by CT, MRI or by blood chemistry tests, dosing of tumor markers and / or molecular biology tests in the case of prostate tumors or hematologic tumors (e.g. PSA in patients affected by prostate cancer, BCR / Abl mRNA in the case of patients undergoing treatment with kinase inhibitors for CML; CM in the case of patients undergoing treatment for multiple myeloma).
* Long-term efficacy (progression-free survival, overall survival).
* Effect of FMD on HOMA index, PCR, circulating levels of IGF-1 and urinary levels of ketone bodies.
* Effect of FMD on lymphocyte subsets, NK cells and antigen-presenting cells with a role documented in antitumor immunity.

It is foreseen that 60 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age > 18 years
* Patients with solid or hematologic tumors undergoing active treatment, including patients who are preparing to start a new treatment with chemotherapeutic regimens, hormone therapies, other molecularly targeted therapies (including kinase inhibitors), biologics (including trastuzumab) , pertuzumab, cetuximab and bevacizumab) or inhibitors of immune checkpoints (eg Opdivo, Keytruda), ie patients in whom treatment is already underway;
* ECOG performance status 0-1
* Adequate organ function
* BMI >21 kg/m2 (with possibility to also enroll patients with 19<BMI<21 based on the judgement of the treating physician)
* Low nutritional risk according to nutritional risk screening (NRS)

Exclusion criteria:

* Diabetes mellitus;
* Previous therapy with IGF-1 inhibitors;
* Food allergies to the components of the FMD;
* BMI <19 kg/m2;
* bio-impedance phase angle <5.0°;
* medium/high nutritional risk according to NRS;
* Any metabolic disorder that can affect gluconeogenesis or ability to adapt to fasting periods;
* Patients who live alone or are not adequately supported by the family context;
* Treatment in progress with other experimental therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
percentage of prescribed diet consumed and intake of any extra food | 6 months
  Feasibility will be monitored through the compilation of a food diary and is defined as the strict adherence to the diet prescribed in all its days with the possibility to admit the consumption of only 50% of the planned diet and / or a maximum consumption of 4- 5 Kcal / kg of food not expected in only one of the days -2, -1, +1 of each cycle.
Quantification of FMD-emergent adverse events | 6 months
  The side effects of Prolon (hematologic and non-hematologic) will be classified according to NCI CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Nencioni, MD, Principal Investigator — Universita degli Studi di Genova
Locations (1):
- Alessio Nencioni, Genoa, GE, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valdemarin F, Caffa I, Persia A, Cremonini AL, Ferrando L, Tagliafico L, Tagliafico A, Guijarro A, Carbone F, Ministrini S, Bertolotto M, Becherini P, Bonfiglio T, Giannotti C, Khalifa A, Ghanem M, Cea M, Sucameli M, Murialdo R, Barbero V, Gradaschi R, Bruzzone F, Borgarelli C, Lambertini M, Vernieri C, Zoppoli G, Longo VD, Montecucco F, Sukkar SG, Nencioni A. Safety and Feasibility of Fasting-Mimicking Diet and Effects on Nutritional Status and Circulating Metabolic and Inflammatory Factors in Cancer Patients Undergoing Active Treatment. Cancers (Basel). 2021 Aug 9;13(16):4013. doi: 10.3390/cancers13164013. PMID 34439167